CLINICAL TRIAL: NCT02863653
Title: Factors Associated With Participation Restrictions in Individuals With Rheumatoid Arthritis
Brief Title: Participation Restrictions in Rheumatoid Arthritis
Status: Completed | Type: Observational
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, Júnia Amorim Andrade, PHD, Federal University of Minas Gerais
Other Study IDs: ETIC 024/09
Record Dates: First submitted 2016-07-20; First posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-07

CONDITIONS: Rheumatoid Arthritis
Keywords: social participation; International Classification of Functioning
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Observation

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: observational study — application of several standard instruments in patients with rheumatoid arthritis

SUMMARY:
Objective: To evaluate what factors contribute to social participation restrictions in subjects with Rheumatoid Arthritis (RA), considering the model International Classification of Functioning (ICF).

Methods: Cross-sectional study with 81 individuals with Rheumatoid Arthritis, using instruments to measure two constructs of component social participation.

DETAILED DESCRIPTION:
In this study the definition of social participation considered several areas, such as marriage and family, work, leisure, religion, economy, and politics which are based in the social scales of the questionnaires SF-36 and AIMS2.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years of age
* Mental capacity as assessed by the Brazilian version of Mini Mental State Examination
* Diagnosis of RA according to the American College of Rheumatology (ACR) 1987 criteria established by attending service rheumatologist.

Exclusion Criteria:

* Individuals who had undergone surgery of the upper limbs, were unable to comply with the protocol for data collection, or with non-corrected visual deficits that could interfere with their functionality were excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For this cross-sectional study involved 81 individuals treated between June 2009 and August 2010 in Clinics Hospital, Universidade Federal de Minas Gerais in Belo Horizonte, Brazil. Recruted by convenience sampling
Sampling Method: Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2009-06; Primary Completion 2009-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
The Short Form Instruments (social aspect) and Arthritis Impact Measurement Scale (social interaction) were used as outcome measures to assess the social participation according to the International Classification of Functioning, Disability and Health | June 2009 to August 2010
  We evaluated 81 individuals in a single meeting with the SF-36 and AIMS2, each participant was assessed for 2 hours. The revised AIMS2 comprises five main dimensions. The score of each AIMS scale varies from zero to 10 (a score of 10 indicates the worst state of health). The SF-36 is a generic instrument that assesses quality of life and comprises eight dimensions. The SF-36 final score varies from zero to 100 in each of the eight dimensions (a score of 100 represents the best state of health).

IPD SHARING:
Plan to Share IPD: No